CLINICAL TRIAL: NCT03264612
Title: Effect of Aeropbic Exercise as Swimming on Premenstrual Syndrome
Brief Title: Effect of Swimming on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise; Swimming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimming group (Active Comparator): Females in group I were instructed to engage into swimming exercise 30 minutes daily, 3 times weekly for 3 months. Exercise was ceased on the first 3 days of menstrual cycle then resumed afterwards.
  The exercise included three stages: warming up, swimming and cooling down.
  Interventions: Behavioral: Aerobic exercise
- Non swimming group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Aerobic exercise — Females in group I were instructed to engage into swimming exercise 30 minutes daily, 3 times weekly for 3 months. Exercise was ceased on the first 3 days of menstrual cycle then resumed afterwards.
  The exercise included three stages: warming up, swimming and cooling down.
  Other Names: Swimming
  Arms: Swimming group

SUMMARY:
Each female sets her experience of 47 manifestations on a 6 point scale separately for the premenstrual, menstrual and intermenstrual phases of her latest and worst menstrual cycle. Daily Symptoms Report was filled at the start and at end of the study (before and after performing swimming exercise) Females in group I were instructed to engage into swimming exercise 30 minutes daily, 3 times weekly for 3 months. Exercise was ceased on the first 3 days of menstrual cycle then resumed afterwards.

The exercise included three stages: warming up, swimming and cooling down.

DETAILED DESCRIPTION:
Each female sets her experience of 47 manifestations on a 6 point scale separately for the premenstrual, menstrual and intermenstrual phases of her latest and worst menstrual cycle. Daily Symptoms Report was filled at the start and at end of the study (before and after performing swimming exercise) Females in group I were instructed to engage into swimming exercise 30 minutes daily, 3 times weekly for 3 months. Exercise was ceased on the first 3 days of menstrual cycle then resumed afterwards.

The exercise included three stages: warming up, swimming and cooling down. Warming up phase involved 5 minutes of breathing, circulatory and stretching exercises. Breathing diaphragmatic and costal exercise was performed. Diaphragmatic breathing exercise was performed at a convenient position with full relaxation, then she inspires deeply through the nose, ballooning her abdomen then expires through the mouth with a sigh and slowly and that was repeated 3-5 times.

Costal breathing exercise was done also at the woman favorable position then she inspires deeply through the nose, opens out her ribs then expires through the mouth with a sigh and slowly and that was repeated 3-5 times..

Circulatory foot and ankle exercises were done by instructing the woman to point her toes up and down, doing isometric calf muscle contractions and knee flexion and extension.

Stretching exercise of neck flexors, extensors, latissimus dorsi, Deltoid dorsal fibers, triceps, pectoralis major, supraspinatus, wrist , lumbar extensors, abdominal, lumbar flexors, lumbar rotators, hamstrings, adductor, gluteal, gastrocnemius, hip flexors, tensor fascia latae and quadriceps muscles were performed during warming up phase.

The second phase of treatment was swimming for 20 minutes starting with 5 minutes walking inside the pool around its edges, then forth and back swimming without reaching fatigue level for 15 minutes.

The last phase was cooling down phase which was the same exercises of the warming up phase for 5 minutes

ELIGIBILITY:
Inclusion Criteria:

1. virgins.
2. Their age ranged from 18 to 25 years old
3. Their body mass index (BMI) ranged from 18 to 25 kg/m2.
4. They were clinically and medically stable during the study
5. Have regular menstrual cycle of 23 to 35 days duration

Exclusion Criteria:

1. cardiopulmonary or orthopaedic problems
2. women taking any hormonal drugs or drugs that affect hormones as antidepressnats during the preceding 3 months before participation in the study
3. any abnormality in ovulation or those with pelvic inflammatory diseases (PID).
4. Women with endocrine abnormality as thyroid, pituitary or ovarian disorders

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2016-04-03 (Actual); Primary Completion 2017-05-14 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Premenstrual distress questionnaire | 3 months after start of swimming
  47 manifestations on a 6 point scale separately for the premenstrual, menstrual and intermenstrual phases of her latest and worst menstrual cycle. Daily Symptoms Report was filled at the start and at end of the study (before and after performing swimming exercise)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Abbassy AH, Sakr HRS, Elsawah H, Wagih H, Ogila AI, Kotb A. Effect of swimming exercise on premenstrual syndrome. Arch Gynecol Obstet. 2018 Apr;297(4):951-959. doi: 10.1007/s00404-018-4664-1. Epub 2018 Jan 19. PMID 29350276